CLINICAL TRIAL: NCT07183332
Title: Comparison of Clinical Effects Between Routine and High-frequency Follow-up After Hemorrhoids Surgery: a Single-center, Prospective, Open-label, Randomized Clinical Trial
Brief Title: Comparison of Clinical Effects Between Routine and High-frequency Follow-up After Hemorrhoids Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PutianU-009
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Follow-up; Quality of Life
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (No Intervention): Patients received routine health education services at discharge and were enrolled in the sample data collection cluster. Patients were followed up by telephone by trained medical and nursing teams at 1 week and 1 month after discharge, and then every 3 months until the end of the one-year follow-up period
- High frequency group (Experimental): Patients received routine health education services at discharge and were enrolled in the sample data collection cluster. Patients were followed up by telephone by a trained medical team at 1, 2, 3, and 4 weeks after discharge, and then every month until the end of the one-year follow-up period.
  Interventions: Behavioral: High frequency follow-up

INTERVENTIONS:
Behavioral: High frequency follow-up — Patients in the high-frequency group received regular follow-ups at a high frequency after discharge.
  Arms: High frequency group

SUMMARY:
This study aims to investigate whether frequent follow-ups can enhance the quality of life of patients after hemorrhoid surgery and reduce the incidence of complications. A total of 116 eligible patients were randomly and evenly divided into two groups (58 patients in each group): A. The control group: Patients received routine health education services upon discharge and were then followed up by phone at the regular frequency. B. The high-frequency group: Patients received routine health education services upon discharge and were then followed up by phone at a higher frequency. The quality of life of the patients and the incidence of complications were compared to evaluate the clinical effects of different intervention measures. The main hypothesis is that compared to conventional care, frequent follow-ups can significantly improve the quality of life of patients, promote wound healing, and reduce the incidence of complications and disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old < age < 75 years old;
* Mixed hemorrhoids were diagnosed;
* Internal hemorrhoids ligation + external hemorrhoidectomy
* Complete hospital records;⑤voluntary cooperation in the study

Exclusion Criteria:

* The patient had mental illness;
* Serious underlying diseases;
* pregnant or lactating women;
* Serious complications and drug allergy occurred during the treatment;
* Communication difficulties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life SCORES | Baseline, weeks 2, 4, 12, 24, 48
  By evaluating the quality of life of patients, we proved the effectiveness of different frequency of follow-up methods in improving the quality of life of patients after hemorrhoids surgery.

SECONDARY OUTCOMES:
pain score | Baseline, Day 7, 14, 21, 28
  The assessment is conducted using the Numerical Rating Scale for Pain (NRS), which requires patients to select an integer (whole number) from 0 to 10 that best describes their pain. 0 typically indicates "no pain", while 10 represents "the most severe pain imaginable".
Complication incidence | Within six months after discharge
  Record the recurrence of hemorrhoids and the occurrence of complications in the patients in the medium and long term. The complications mainly include: incision infection, wound bleeding, and urinary retention.
patient satisfaction | Baseline, weeks 2, 4, 12, 24, 48
  The Patient Satisfaction Questionnaire Short Form (PSQ-18) was used for measurement during the telephone follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Putian University Affiliated Hospital, Putian, China

IPD SHARING:
Plan to Share IPD: No
Based on a strict commitment to participant privacy protection, compliance with the terms of the ethical review protocol, and adherence to the sponsoring institution's policies, IPD from this study will not be shared at this time.